CLINICAL TRIAL: NCT00297193
Title: Autologous Stem Cell Transplantation for Crohn's Disease: ASTIC
Brief Title: ASTIC Autologous Stem Cell Transplantation for Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For safety reasons the recruitment was halted prematurely. Patients on the trial continute to receive treatment and are being followed up as part the protocol.
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: The Broad Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT2005-003337-40; ASTIC
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2013-08

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; HSCT; Autologous; EBMT; ECCO
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant Arm (Experimental): Hematopoietic stem cell mobilisation followed, within 4 weeks, by high dose immunoablation and autologous stem cell transplantation
  Interventions: Procedure: Autologous haematopoietic stem cell transplant
- Delayed Transplant (Experimental): Hematopoietic stem cell mobilisation followed, after 59 weeks, by high dose immunoablation and autologous hematopoietic stem cell transplantation
  Interventions: Procedure: Autologous haematopoietic stem cell transplant

INTERVENTIONS:
Procedure: Autologous haematopoietic stem cell transplant — All patients will be mobilised prior to randomisation. Those receiving early transplantation will be compared over the first year with those whose transplant has been delayed.

SUMMARY:
Transplant study for patients with relapsing Crohn's disease demonstrating clear intolerance or toxicity to conventional treatment.

The purpose of this study is to determine whether there is a potential clinical benefit of hematopoietic stem cell mobilisation followed by high dose immuno-ablation and autologous stem cell transplantation versus hematopoietic stem cell mobilisation only followed by best clinical practice.

DETAILED DESCRIPTION:
Open label, phase III, randomised, multicentre study comparing early transplantation procedure with transplantation carried out to the same protocol but delayed by one year. The status of patients undergoing early HSCT will be evaluated after one year and compared to those about to undergo delayed HSCT

Patients will be randomised to:

* Hematopoietic stem cell mobilisation followed, within 4 weeks, by high dose immunoablation and autologous stem cell transplantation
* Hematopoietic stem cell mobilisation followed, after 59 weeks, by high dose immunoablation and autologous hematopoietic stem cell transplantation

All patients will be mobilised prior to randomisation. Those receiving early transplantation will be compared over the first year with those whose transplant has been delayed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria: mandatory

1. Age between 18 and 50 years (Patients aged 50-65 can participate if specially approved by the Trial Steering Committee)
2. Confirmed diagnosis of active Crohn's Disease
3. Unsatisfactory course despite 3 immunosuppressive agents (usually azathioprine, methotrexate and infliximab) in addition to corticosteroids. Patients should have relapsing disease (i.e. >1 exacerbation/year) despite thiopurines, methotrexate and/or infliximab maintenance therapy or clear demonstration of intolerance / toxicity to these drugs.
4. Impaired function and quality of life, compared to population means, on at least one of the following:

   1. IBDQ (Appendix 6)
   2. European Questionnaire of Life quality (EuroQOL-5D, Appendix 4)
   3. Impaired function on Karnofsky index (Appendix 7)
5. Current problems unsuitable for surgery and patient at risk for developing short bowel syndrome.
6. Informed consent

Inclusion criteria: discretionary

1. Wherever possible, diseased tissue should be accessible endoscopically for objective histological study but in the case of small bowel disease that is extensive but does not extend to duodenum or terminal ileum, participation without endoscopy is allowed.
2. Smokers may enter the study provided they have received intensive counselling about smoking.
3. Add patients with ileostomy/colostomy and patients with short bowel syndrome

Exclusion Criteria:

1. Pregnancy or unwillingness to use adequate contraception during the study
2. Concomitant severe disease
3. Diarrhoea due to short small or large bowel
4. Infection or risk thereof
5. Significant malnutrition: Body Mass Index (BMI) ≤18, serum albumin <20 g/l
6. Previous poor compliance
7. Concurrent enrolment in any other protocol using an investigational drug or hematopoietic growth factor up to four weeks before study entry.
8. Lack of funding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-06; Primary Completion 2013-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Proportion patients in sustained disease remission | 1 year
  To evaluate the potential clinical benefit of hematopoietic stem cell mobilisation followed by high dose immuno-ablation and autologous stem cell transplantation versus hematopoietic stem cell mobilisation only followed by best clinical practice in patients with Crohn' s disease.

SECONDARY OUTCOMES:
patients who have not responded to immunosuppressant medication | 1 - 2 years
  To evaluate the safety of Hematopoietic Stem Cell Transplantation (HSCT) in Crohn's disease patients who have not responded to immunosuppressant medication

OTHER OUTCOMES:
Impact of HSCT on health related, and generic, quality of life measures | 1 - 2 Years
  To evaluate the impact of HSCT on health related, and generic, quality of life measures
To identify factors predictive of success | 1-2 years
  To identify factors predictive of success

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hawkey, Study Chair — Nottingham University Hospital - Wolfson Digestive Diseases Centre
Locations (19):
- University Hospital Gasthuisberg, Leuven, Herestraat 49, Belgium
- University of Calgery, Calgary, Alberta, Canada
- France (2):
  - Hopital Huriez Chru, Lille
  - Hospital Sanin-Louis, Paris
- Italy (7):
  - Dipatimento di Medicina Interna E Gastroenterologia, Bologna
  - Universita di Bologna Interna e Gastroenterologia Policlinico Saint Orsola, Bologna
  - Careggi Hospital, Florence
  - Istituto Clinico Humanitas, Milan
  - Fondazione IRCCS Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Milan
  - L Sacco University Hopsital, Milan
  - Casa Sollievo Della Sofferenza IRCCS Hospital, San Giovanni Rotondo
- Hospital Universitari Germans Trias I Pujol, Dept of Gastroenterology, Badalona, Spain
- Switzerland (2):
  - University Hospital, Basel
  - Universitätsspital Zürich, Zurich
- United Kingdom (5):
  - The John Radcliffe Hospital, Oxford, Headington
  - Western General Hospital, Edinburgh
  - Barts and the London NHS Trust, London
  - City Hospital, Nottingham
  - Nottingham Digestive Diseases Centre, Nottingham

REFERENCES:
- [Derived] Lindsay JO, Allez M, Clark M, Labopin M, Ricart E, Rogler G, Rovira M, Satsangi J, Farge D, Hawkey CJ; ASTIC trial group; European Society for Blood and Marrow Transplantation Autoimmune Disease Working Party; European Crohn's and Colitis Organisation. Autologous stem-cell transplantation in treatment-refractory Crohn's disease: an analysis of pooled data from the ASTIC trial. Lancet Gastroenterol Hepatol. 2017 Jun;2(6):399-406. doi: 10.1016/S2468-1253(17)30056-0. Epub 2017 Apr 6. PMID 28497755
- [Derived] Hawkey CJ, Allez M, Clark MM, Labopin M, Lindsay JO, Ricart E, Rogler G, Rovira M, Satsangi J, Danese S, Russell N, Gribben J, Johnson P, Larghero J, Thieblemont C, Ardizzone S, Dierickx D, Ibatici A, Littlewood T, Onida F, Schanz U, Vermeire S, Colombel JF, Jouet JP, Clark E, Saccardi R, Tyndall A, Travis S, Farge D. Autologous Hematopoetic Stem Cell Transplantation for Refractory Crohn Disease: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2524-34. doi: 10.1001/jama.2015.16700. PMID 26670970